CLINICAL TRIAL: NCT00525876
Title: Allogeneic Stem Cell Transplantation With Rituximab Containing Nonablative Conditioning Regimen for Advanced/Recurrent Mantle Cell Lymphoma
Brief Title: Non-Myeloablative Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0309
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Results first posted 2011-12-07 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-11

CONDITIONS: Lymphoma
Keywords: Mantle Cell Lymphoma; Lymphoma; Allogeneic Stem Cell Transplant; Rituximab; Cyclophosphamide; Neosar; Cytoxan; Fludarabine; Fludara; Fludarabine phosphate; Rituxan; Alemtuzumab; CAMPATH-1H; Campath; Total Body Irradiation; TBI
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Rituximab; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Matched Sibling Transplant (Experimental): Allogeneic Stem Cell Transplantation With Rituximab Containing Nonablative Conditioning Regimen: Cyclophosphamide 750 mg/m^2 given intravenously on Day -3, 4 hours after completion of Fludarabine 30 mg/m^2 given intravenously on Days -5 and -3 before transplantation. Rituximab 375 mg/m^2 given intravenously on Days -13, -6 before transplantation and Days 16, 8 after transplantation.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rituximab; Procedure: Allogeneic Stem Cell Infusion
- Allo MUD & MM (Experimental): Allo MUD & MM = Allogeneic Stem Cell Transplantation, Matched unrelated donor or mismatched sibling donor transplantations: Cyclophosphamide 1000 mg/m^2 given intravenously on Day -3, 4 hours after completion of Fludarabine 30 mg/m^2 given intravenously on Days -5 and -3 before transplantation. Rituximab 375 mg/m^2 given intravenously on Days -8, -1 before transplantation and Days 6, 13 after transplantation. Alemtuzumab 15 mg per day given intravenously days 1 through 3 after transplantation.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rituximab; Drug: Alemtuzumab; Procedure: Allogeneic Stem Cell Infusion

INTERVENTIONS:
Drug: Cyclophosphamide — Matched Donors:
  750 mg/m^2 given intravenously on Day -3, 4 hours after completion of Fludarabine.
  Unrelated or Mismatched Donors:
  1000 mg/m^2 given intravenously on Day -3, 4 hours after completion of Fludarabine.
  (Stem Cell Transplantation and Low Dose Total Body Irradiation = Day 0)
  Other Names: Cytoxan; Neosar
Drug: Fludarabine — 30 mg/m^2 given intravenously on Days -5 and -3 before transplantation.
  (Stem Cell Transplantation and Low Dose Total Body Irradiation = Day 0)
  Other Names: Fludarabine phosphate; Fludara
Drug: Rituximab — Matched Donors:
  375 mg/m^2 given intravenously on Days -13, -6 before transplantation and Days 16, 8 after transplantation.
  Unrelated/Mismatched Donors:
  375 mg/m^2 given intravenously on Days -8, -1 before transplantation and Days 6, 13 after transplantation.
  (Stem Cell Transplantation and Low Dose Total Body Irradiation = Day 0)
  For development of disease progression or no response, immunomanipulation with Rituximab 375 mg/m^2 given intravenously, then 1000 mg/m^2 given intravenously weekly for 3 weeks, and taper off Tacrolimus dose over 2 weeks.
  DLI = Donor Lymphocyte Infusion/Immunomodulation Post Transplantation Immunomodulation for patients with lymphoid Malignancies:
  375 mg/m^2 then 1000 mg/m^2 weekly x 3 if immunomanipulation is undertaken for persistent disease.
  Other Names: Rituxan
Drug: Alemtuzumab — Unrelated/Mismatched Donors:
  15 mg per day given intravenously days 1 through 3 after transplantation.
  (Stem Cell Transplantation and Low Dose Total Body Irradiation = Day 0)
  Other Names: CAMPATH-1H; Campath
  Arms: Allo MUD & MM
Procedure: Allogeneic Stem Cell Infusion — Infusion of stem cells.
  Other Names: ASCT

SUMMARY:
1. To determine the safety and efficacy of non-myeloablative allogeneic stem cell transplantation using rituximab, cyclophosphamide, fludarabine as a preparative regimen for patients with advanced or recurrent mantle cell lymphoma.
2. To determine factors associated with response and durable remission in patients receiving rituximab, cyclophosphamide, and fludarabine in preparation for allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
MATCHED SIBLING TRANSPLANTS:

If you are found to be eligible to take part in this study, you will be admitted to the hospital to receive treatment. Two (2) chemotherapy drugs, fludarabine and cyclophosphamide, will be given each day for 3 days. The drugs will be given one at a time in a vein. Each treatment will take about 30 minutes. Fludarabine will be given first, and cyclophosphamide will be given 4 hours later. You will receive rituximab once a week for 4 weeks by vein over 4-8 hours. The first dose will starts one week before starting the chemotherapy.

Two days after finishing chemotherapy, you will receive a transplant of stem cells from a sibling. The stem cells will be infused into your vein. Seven days later, you will begin to receive a drug called granulocyte colony-stimulating factor (G-CSF). G-CSF helps the new stem cells do their normal work in the body;making new blood cells. You will receive G-CSF each day until your blood cell counts begin to recover to a certain level.

Sometimes the donor cells cause inflammation of the skin, liver and gut, and a reaction called graft-versus-host disease occurs. The drugs tacrolimus and methotrexate will be given to help decrease the risk of this. These drugs are also given through a vein before and after transplant . Tacrolimus will be infused two days before transplant and will continue to be given daily as a continuous infusion. Methotrexate will be given through the vein as a short infusion on Days 1, 3, and 6 after the transplant. Tacrolimus also comes in pill form, and you may switch to the pills when ready.

During your hospitalization, you will be examined daily, and blood (about 1 tablespoon) samples will be taken daily to evaluate your blood count levels, the function of your liver and kidneys, as well as electrolytes. This blood will also be used to measure tacrolimus levels and to look for any infections. You might be given blood transfusions if blood cell counts remain low.

MATCHED UNRELATED OR MISMATCHED SIBLING TRANSPLANTS:

Alemtuzumab is a drug that is designed to specifically attack some types of leukemia and lymphoma cells. In addition, it weakens the immune system, helping to prevent the rejection of donor marrow or stem cells.

TBI is designed to damage the DNA (the genetic material of cells) of cancer cells, which may kill the cancer cells.

Cyclophosphamide is designed to interfere with the multiplication of cancer cells, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

Fludarabine is designed to make cancer cells less able to repair damaged DNA. This may increase the likelihood of the cells dying.

Rituximab is designed to attach to lymphoma cells, which may cause them to die.

If you are found to be eligible to take part in this study, you will be admitted to the hospital for treatment. Alemtuzumab will be injected into your vein over a period of 4 hours. This will be done 3 days in a row (Days 1 to 3). Drugs diphenhydramine (Benadryl), solumedrol and acetaminophen (Tylenol) will be given in to decrease the risk of or ease side effects before each dose of the alemtuzumab.

You will also receive fludarabine and cyclophosphamide once a day for 3 days. They will be given on the same days as alemtuzumab. Both drugs will be given through a catheter (plastic tube) that extends into the large chest vein. The catheter will be left in place throughout treatment on this study. Some participants, depending on their type of disease, will also receive rituximab. Rituximab will be given 8 days before the transplant and then once a week for a total of 4 doses.

After completion of chemotherapy, you will receive TBI, and later on the same day, blood stem cells from a donor will be given through the catheter. G-CSF, a growth factor that promotes the production of blood cells, will be injected under the skin once a day until your blood cell counts recover to a certain level.

Blood tests (about 2 tablespoons each) , urine tests, bone marrow aspirations, and x-rays will be done as needed to track the effects of the transplant. The blood tests will be drawn daily while in the hospital and then at least twice weekly as an outpatient for the first 100 days. The CT scans and bone marrow studies will be done at 1, 3, 6, and 12 months and then every 6 months for at least 3 years after transplant. You may also have transfusions of blood and platelets as needed.

IMMUNOMODULATION POST NONABLATIVE STEM CELL TRANSPLANTATION FOR PATIENTS WITH LYMPHOID MALIGNANCIES:

You will receive treatment as an outpatient. You will receive rituximab over 4 - 8 hours through a vein once a week for 4 weeks. You will also get a boost of cells from the same donor from whom you received the original transplant. These additional cells will be infused through the vein (over 30 - 60 minutes) between the second and the third dose of rituximab. The infusion may have to be done later if cells were not available as scheduled.

Sometimes the donor cells cause inflammation of the skin, liver and gut, and a reaction called graft-versus-host disease occurs. If this happens, the drug tacrolimus and methotrexate will be given to help control this reaction. These medications are usually given by pills on a daily basis.

A boost with a higher number of cells may be infused once a month for 3 months if there is no graft-versus-host disease and if disease remains.

During treatment, you will be examined as needed, and blood samples (1 tablespoon once or twice a week) will be taken for routine tests. You may need to receive blood transfusions during this study if your blood cell counts remain low.

******

About 40 patients will take part in this study, and all will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients can be as old as 70 years.
2. They must have a diagnosis of MCL, either (1) Recurrent, (2) Newly diagnosed (after cytoreduction with conventional chemotherapy) but with high-risk features (blastic or blastoid features, leukemic phase, or elevated B^2 microglobulin (> 3).
3. Patients that have received prior conventional chemotherapy but have not achieved complete response (CR).
4. Disease must be chemosensitive, (ie, patients must not have had a partial response to prior therapy).
5. Patients whose disease failed to respond to a previous autologous transplantation may also be eligible.
6. Patients must have a matched or 1 antigen mismatched sibling or unrelated donor.
7. Point Scale (PS) </= 2.
8. Inclusion criteria for Immunomodulation Post transplantation: Patients can be as old as 70 years. Patients must have a diagnosis of MCL or CLL with one of the following characteristics: 1. Patients who develop disease progression or do not experience a CR within 3 months post-allogeneic transplantation 2. Patients with a weak chimerism (any mixed chimerism of donor T cells in patients receiving Campath by day 90, and less than 20% for patients not receiving Campath) or a drop of 20% or more with an amount of donor cells present in the blood < 50% by PCR .
9. Continued from Inclusion # 8: Patients must have the same donor of the original transplant willing to donate lymphocytes. 4. PS </ 2.

Exclusion Criteria:

1. Past history of anaphylaxis following exposure to rat- or mouse-derived CDR-grafted humanized monoclonal antibodies.
2. Less than 4 weeks since prior chemotherapy counted from first day of treatment regimen.
3. Pregnancy or lactation.
4. HIV or HTLV-I positivity.
5. Serum creatinine concentration > 1.6 mg/dl or serum bilirubin > 2.0 mg/dl unless due to tumor
6. pulmonary function test - carbon monoxide diffusing capacity < 40%
7. cardiac ejection fraction < 40% of predicted levels (by multiple-gated acquisition or echocardiography).
8. Severe concomitant medical or psychiatric illness.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa F. Khouri, MD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period:1/27/2005 through 8/31/2010. All participant recruitment attempted at UT MD Anderson Cancer Center.
Pre-assignment Details: Out of the 49 participants enrolled, 13 were excluded, not assigned to part of the two intervention study groups.
Period: Overall Study
Arm/Group | Matched Sibling Transplant | Allo MUD & MM
Started | 16 | 20
Completed | 16 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Matched Sibling Transplant | Allo MUD & MM | Total
Number analyzed (Participants) | 16 | 20 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (7) | 59 (6) | 59 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 9 | 16 | 25
Region of Enrollment [Number; unit: participants]
  United States | 16 | 20 | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 100 Days Post Transplant (Number of Surviving Participants)
Description: Overall Survival defined as the number of participants living at day 100 following non-myeloablative allogeneic stem cell transplantation using rituximab, cyclophosphamide, fludarabine as a preparative regimen for participants with advanced or recurrent mantle cell lymphoma.
Time Frame: 100 days post transplant
Population: Analysis was per protocol.
Measure: Number; unit: participants
Arm/Group | Matched Sibling Transplant | Allo MUD & MM
Number analyzed (Participants) | 16 | 20
participants | 16 | 19

ADVERSE EVENTS:
Time Frame: 3 years and 3 months
Arm/Group | Matched Sibling Transplant | Allo MUD & MM
Serious Adverse Events (participants affected / at risk) | 3/16 | 2/20
Other Adverse Events (participants affected / at risk) | 15/16 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matched Sibling Transplant (N=16) | Allo MUD & MM (N=20)
Allergic Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Tongue swelling
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Aspergillus Infection (Infections and infestations) | 1 (1) | 0 (0)
Prolonged Hospitalization due to Graft vs Host Disease (General disorders) | 1 (1) | 0 (0)
CMV Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Matched Sibling Transplant (N=16) | Allo MUD & MM (N=20)
Epistaxis (General disorders) | 0 (0) | 1 (1)
Lower Extremity Edema (Cardiac disorders) | 1 (1) | 3 (3)
Decreased Left Ventricular Ejection Fraction (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 5 (5) | 6 (6)
Hypotension (Cardiac disorders) | 4 (4) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 7 (7) | 8 (8)
Chills (General disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 3 (3)
Mucositis (Gastrointestinal disorders) | 3 (3) | 5 (5)
Lower GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (12) | 15 (15)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Elevated Creatinine (Renal and urinary disorders) | 3 (3) | 7 (7)
Hemorrhagic Cystitis (Renal and urinary disorders) | 3 (3) | 5 (5)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Elevated Alkaline Phosphatase (Hepatobiliary disorders) | 5 (5) | 10 (10)
Elevated Alanine Aminotransferase (Hepatobiliary disorders) | 6 (6) | 6 (6)
Elevated Bilirubin (Hepatobiliary disorders) | 3 (3) | 1 (1)
Confusion (Nervous system disorders) | 1 (1) | 2 (2)
Headache (General disorders) | 6 (6) | 4 (4)
Hearing Loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 3 (3) | 3 (3)
CNS Hemorrhage (General disorders) | 1 (1) | 0 (0)
Bone Pain (General disorders) | 4 (4) | 3 (3)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 13 (13)
Graft versus Host Disease (General disorders) | 6 (6) | 3 (3)
Infections (Infections and infestations) | 11/11 (11) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes